CLINICAL TRIAL: NCT04165135
Title: A Multicenter, Non-Interventional Study to Evaluate Physical Activity, Bleeding Incidence and Health Related Quality of Life, in Patients With Haemophilia A Without Inhibitors Receiving Standard of Care Treatment
Brief Title: An Observational Study to Evaluate Physical Activity, Bleeding Incidence and Health Related Quality of Life, in Participants With Haemophilia A Without Inhibitors Receiving Standard of Care Treatment
Acronym: POWER
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML40983
Record Dates: First submitted 2019-10-31; First posted 2019-11-15 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-01

CONDITIONS: Severe Hereditary Factor VIII Deficiency Disease Without Inhibitor; Moderate Hereditary Factor VIII Deficiency Disease Without Inhibitor; Haemophilia A
Keywords: Hemophilia A; Factor VIII
MeSH Terms: conditions — Hemophilia A | interventions — Standard of Care; Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Haemophilia A Without FVIII Inhibitors
  Interventions: Drug: Standard of Care for Haemophilia A

INTERVENTIONS:
Drug: Standard of Care for Haemophilia A — There is no pre-determined studied medicinal product. Any treatment (including treatments started during the observational period) will be administered according to standard clinical practice, independently of participation in the current study, according to clinician's independent therapeutic decision.

SUMMARY:
This multicenter, non-interventional, prospective study will collect information about activity status, bleeds, health-related quality of life (HRQoL), health status, and safety in participants with moderate or severe haemophilia A without factor VIII (FVIII) inhibitors, who are being treated in accordance with normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Must own a device compatible with the electronic Patient-Reported Outcome (ePRO) application and with the fitness tracker that will be provided to the patient
* Must have on his/her own device a data traffic availability of at least 2 gigabytes (GB) in total per month intended only for use of study applications and data transfer. If the data traffic plan is exhausted, the participant must be able to connect to a wi-fi network at least once every day in order to transfer the data collected for the study purpose
* Must accept to run on his/her own device the ePRO application and the fitness tracker application
* Must be available to turn on daily the bluetooth connection of his/her own device in order to allow the synchronization with the fitness tracker
* Ability and willingness to comply with all aspects of the protocol, including completion of questions on the ePRO application (for underage population, ePRO questions can be answered by legally authorized representative if deemed necessary)
* Ability and willingness to wear the activity tracking device as indicated
* Diagnosis of severe (FVIII <1%) or moderate (FVIII ≥1% and ≤2%) congenital haemophilia A
* No prior history of a positive inhibitor against FVIII. If participant has a previous history of inhibitor development, the participant must have successfully eradicated inhibitors since 3 years.
* At least 150 exposure days of FVIII prior to enrolment

Exclusion Criteria:

* Bleeding disorder other than congenital haemophilia A
* Ongoing (or planned during the study) immune tolerance induction or FVIII prophylaxis if the participant has currently low titre of inhibitors or had inhibitors in the past 3 years
* Previous or concomitant autoimmune or connective tissue disease
* History of or suspected allergy or intolerance to any of the component of the fitness device (e.g., aluminium anodised)
* History of clinically significant hypersensitivity associated with monoclonal antibody
* Obesity (Body Mass Index [BMI] ≥30 kilograms/metre squared of body surface area [kg/m^2})
* Clinically important cardiovascular, metabolic, endocrine disorders or any other concomitant diseases or conditions that could limit the mobility of participant or could represent any risk according to the Investigator's judgment, or that could interfere with the study evaluation parameters
* Participation in any other interventional clinical trial, including Roche sponsored studies or in any other support program that may include drug administration other than standard clinical practice (e.g., compassionate use, use not in agreement with the authorized indications, patient support programs, etc.)

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Approximately 150 participants overall, 125 with severe haemophilia A and 25 with moderate haemophilia A without inhibitors against factor VIII (FVIII), are planned to be enrolled at sites across Italy.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Italy (17):
  - AOU Cons. Policlinico Bari; Centro Emofilia e Trombosi - UO Medicina Trasfusionale, Bari, Apulia
  - Az. Osp. Pugliese Ciaccio; S. C. Emofilia, Emostasi e Trombosi, Catanzaro, Calabria
  - AOU Federico II; Medicina Clinica Chirurgia Centro Emocoaugulopatie e Emofilia, Napoli, Campania
  - PO Cesena - Osp M. Bufalini; Patologia Clinica - S.S.A. Serv. Medicina Trasf.- Centro Emofilia, Cesena, Emilia-Romagna
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia; Dip Biot Cel e Ematol, Rome, Lazio
  - Ospedale Pediatrico Bambino Gesù; Oncoematologia Centro Emostasi e Trombosi, Rome, Lazio
  - Policlinico Univ. A. Gemelli; Polo di Scienze Oncologiche ed Ematologiche, Rome, Lazio
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico; Centro Emofilia e Trombosi "Angelo Bianchi e Bonomi", Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo; S.C. Medicina Generale 2 - Centro Emofilia, Pavia, Lombardy
  - A.O.Santi Antonio e Biagio e Cesare Arrigo; S.S. Emostasi e Trombosi - Dip. Onco-Ema e Med Spec., Alessandria, Piedmont
  - AO Città Salute e Scienza D-Osp S. G. Battista Molinette; SSCVD Malattie Tromboti e Emorragiche, Turin, Piedmont
  - Osp. Infant. Regina Margherita; S.S.D. Medicina Trasfusionale Materno-infantile Traumatologica, Turin, Piedmont
  - Azienda Uni Ria Policlinico P. Giaccone ; Divisione Di Ematologia E Trapianto, Palermo, Sicily
  - Ospedale Ferrarotto; Divisione Di Ematologia, Via S. Sofia 78, Sicily
  - AOU Careggi; SOD Malattie Emorragiche, Florence, Tuscany
  - Azienda Ospedaliera di Padova; Centro Emofilia, Padua, Veneto
  - Ospedale Di Vicenza; Nefrologia, Ematologia, Vicenza, Veneto

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Petracca F, Tempre R, Cucciniello M, Ciani O, Pompeo E, Sannino L, Lovato V, Castaman G, Ghirardini A, Tarricone R. An Electronic Patient-Reported Outcome Mobile App for Data Collection in Type A Hemophilia: Design and Usability Study. JMIR Form Res. 2021 Dec 1;5(12):e25071. doi: 10.2196/25071. PMID 34855619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 107 patients were screened, but 4 patients did not meet the eligibility criteria; in total, 103 participants were enrolled and started the study. Participants took part in this study at 17 investigative sites in Italy from 24 February 2020 up to 28 April 2022.
Groups:
- Standard of Care for Haemophilia A: Participants with severe or moderate Haemophilia A without inhibitors against Factor VIII, receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Period: Overall Study
Arm/Group | Standard of Care for Haemophilia A
Started | 103
Completed | 88
Not Completed | 15
Not completed — Protocol Violation | 10
Not completed — Participants withdrawal of consent | 5

BASELINE CHARACTERISTICS:
Population: Intention-To-Treat (ITT) population included all enrolled participants who received the electronic patient-reported outcome (ePRO) application and the fitness tracker.
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 93
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 99
  Asian | 2
  American Indian or Alaska Native | 1
  Other | 1
Is Haemophilia A diagnosis confirmed [Count of Participants; unit: Participants]
  Yes | 103
  No | 0
Severity type [Count of Participants; unit: Participants]
  Moderate Haemophilia | 6
  Severe Haemophilia | 97

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Daily Active Minutes of Physical Activity Performed by Participants (by Age Categories: 12-17, 18-30, and 31-50 Years) Over the Course of the Study
Description: Physical activity data was collected as daily active minutes measured on each valid day by wearing a fitness tracker continuously during study participation. Valid day = a day in which fitness tracker was worn for at least 10 hours. Daily active minutes were saved in two different sets of data collected by fitness tracker. For each set minutes were categorized by intensity of activity done. First set = minutes categorized according to time collected in each heart zone. Overall heart zone minutes = fat-burn minutes (heart rate: 50-69% of maximum) + cardio minutes (medium-to-high intensity exercise zone corresponds to heart rate: 70-84% of maximum) + peak minutes (high-intensity exercise zone, corresponds to heart rate > 85% of maximum). Second set =minutes categorized according to active zones. Overall active zone minutes=lightly active minutes +fairly active minutes+very active minutes. Moderate-to-Vigorous Physical Activity (MVPA) minutes=Fairly active minutes+Very active minutes.
Time Frame: From baseline to study completion (up to 18 months)
Population: Evaluable population included all enrolled participants with at least 6 valid months of physical activity evaluations during the study.
Measure: Mean (95% Confidence Interval); unit: number of daily active minutes
Groups:
- Standard of Care: 12-17 Years: Participants who were 12-17 years of age with severe or moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
- Standard of Care: 18-30 Years: Participants who were 18-30 years of age with severe or moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
- Standard of Care:31-50 Years: Participants who were 31-50 years of age with severe or moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care:31-50 Years
Number analyzed (Participants) | 6 | 22 | 26
number of daily active minutes
  Heart Zone Minutes | 53.2 [-45.2 to 151.6] | 24.6 [10.9 to 38.3] | 39.2 [13.9 to 64.6]
  Active Zone Minutes | 226.5 [173.8 to 279.2] | 309.4 [264.6 to 354.1] | 284.1 [246.3 to 321.9]
  MVPA Minutes | 13.8 [0.4 to 27.2] | 42.3 [23.5 to 61.0] | 28.6 [14.2 to 43.0]
Statistical Analysis 1: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Heart zone minutes: Comparison among the age groups was performed by means of a Kruskal-Wallis test; Test type: Other; p = 0.7630, Kruskal-Wallis
Statistical Analysis 2: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Active zone minutes: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.0913, Kruskal-Wallis
Statistical Analysis 3: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; MVPA minutes: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.0956, Kruskal-Wallis

2. Primary Outcome: Mean Number of Steps Taken Per Day by Participants (by Age Categories: 12-17, 18-30, and 31-50 Years) Over the Course of the Study
Description: Number of steps taken by the participants on each valid day were measured by wearing a fitness tracker continuously during study participation. Valid day was defined as a day in which fitness tracker was worn for at least 10 hours.
Time Frame: From baseline to study completion (up to 18 months)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of steps per day
Groups:
- Standard of Care: 31- 50 Years: Participants who were 31-50 years of age with severe or moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care: 31- 50 Years
Number analyzed (Participants) | 6 | 22 | 26
number of steps per day | 5402.4 [3150.3 to 7654.5] | 8788.3 [7233.9 to 10342.7] | 8279.8 [6419.9 to 10139.7]
Statistical Analysis 1: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31- 50 Years; Test type: Other; p = 0.0649, Kruskal-Wallis

3. Primary Outcome: Mean Metabolic Equivalent of Tasks (METs) Per Day Performed by Participants (by Age Categories: 12-17, 18-30, and 31-50 Years) Over the Course of the Study
Description: The MET is an objective measure of the ratio of the rate at which a person expends energy, relative to the mass of that person, while performing some specific physical activity compared to a reference. The METs were derived as: (amount of kilo calories (kcal) collected in the fat-burn, cardio, and peak minutes) / [(sum of fat-burn, cardio and peak hours) * weight of the participant in kilograms (kg)].
Time Frame: From baseline to study completion (up to 18 months)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: MET per day
Groups:
- Standard of Care: 31- 50 Years: Participants who were 31- 50 years of age with severe or moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care: 31- 50 Years
Number analyzed (Participants) | 6 | 22 | 26
MET per day | 5.1 [3.7 to 6.5] | 5.3 [5.1 to 5.5] | 4.5 [4.1 to 4.9]
Statistical Analysis 1: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31- 50 Years; Test type: Other; p = 0.0026, Kruskal-Wallis

4. Secondary Outcome: Mean Rate of the Number of Times Engaging in Physical Activity Per Week by Type of Physical Activity Performed by Participants (by Age Categories: 12-17, 18-30, and 31-50 Years) Over the Course of the Study
Description: The activity weekly rate was derived on a per participant basis as ratio between the number of times that the type of activity is reported on the fitness tracker (numerator) and the length of the observational period (i.e. end of study date - baseline date + 1) (denominator) and then multiplied by 7. The physical activities were categorized in the following groups: exercises at intervals, gym weights, running, swimming, tapis roulant, walk, general exercises: other types of physical activity identified by the fitness tracker that are not already included in the above-mentioned categories.
Time Frame: From baseline to study completion (up to 18 months)
Population: Evaluable population included all enrolled participants with at least 6 valid months of physical activity evaluations during the study. Number analyzed is the number of participants with data available for analysis.
Measure: Mean (95% Confidence Interval); unit: number of times per week
Groups:
- Standard of Care: 31-50 Years: Participants who were 31-50 years of age with severe or moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care: 31-50 Years
Number analyzed (Participants) | 6 | 22 | 26
number of times per week
  Running: number analyzed (Participants) | 5 | 11 | 8
  Running | 0.06 [0.02 to 0.10] | 0.12 [-0.02 to 0.26] | 0.18 [-0.01 to 0.37]
  Swimming: number analyzed (Participants) | 3 | 7 | 8
  Swimming | 0.03 [0 to 0.06] | 0.06 [0.00 to 0.12] | 0.03 [0.02 to 0.04]
  Tapis Roulant: number analyzed (Participants) | 2 | 5 | 3
  Tapis Roulant | 0.06 [0.04 to 0.07] | 0.11 [0.00 to 0.23] | 0.05 [0.02 to 0.08]
  Gym Weights: number analyzed (Participants) | 3 | 3 | 5
  Gym Weights | 0.03 [0.00 to 0.06] | 0.63 [-1.93 to 3.20] | 0.13 [0.03 to 0.23]
  Exercises at Intervals: number analyzed (Participants) | 4 | 6 | 7
  Exercises at Intervals | 0.02 [0.01 to 0.04] | 0.02 [0.01 to 0.04] | 0.02 [0.01 to 0.03]
  General: number analyzed (Participants) | 6 | 22 | 24
  General | 0.86 [0.47 to 1.24] | 0.86 [0.44 to 1.28] | 0.51 [0.34 to 0.68]
  Walk | 0.53 [0.05 to 1.01] | 1.30 [0.97 to 1.63] | 0.88 [0.44 to 1.33]
Statistical Analysis 1: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Running: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.9493, Kruskal-Wallis
Statistical Analysis 2: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Swimming: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.8305, Kruskal-Wallis
Statistical Analysis 3: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Tapis Roulant: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.8725, Kruskal-Wallis
Statistical Analysis 4: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Gym Weights: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.3380, Kruskal-Wallis
Statistical Analysis 5: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Exercises at Intervals: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.9706, Kruskal-Wallis
Statistical Analysis 6: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; General: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.1727, Kruskal-Wallis
Statistical Analysis 7: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Walk: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.0099, Kruskal-Wallis

5. Secondary Outcome: Mean Active Minutes by Intensity (Lightly Active Minutes) for Each Type of Physical Activity Performed by Participants (by Age Categories: 12-17, 18-30, and 31-50 Years) Over the Course of the Study
Description: The number of active minutes by intensity (lightly, fairly, and very active minutes) were obtained at the participant level on a per activity basis as the median of the values collected by the fitness tracker for each activity recorded during the observational period. In this analysis, the means and 95% confidence intervals were calculated using the median lightly active minutes by type of physical activity performed by participants with available data. The physical activities were categorized in the following groups: exercises at intervals, gym weights, running, swimming, tapis roulant, walk, general exercises: other types of physical activity identified by the fitness tracker that are not already included in the above-mentioned categories.
Time Frame: From baseline to study completion (up to 18 months)
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: lightly active minutes per activity
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care:31-50 Years
Number analyzed (Participants) | 6 | 22 | 26
lightly active minutes per activity
  Running: number analyzed (Participants) | 5 | 11 | 8
  Running | 0.1 [-0.2 to 0.4] | 0.5 [0.0 to 1.1] | 0.3 [-0.1 to 0.6]
  Swimming: number analyzed (Participants) | 3 | 7 | 8
  Swimming | 2.7 [-6.7 to 12.1] | 2.8 [0.6 to 5.0] | 3.8 [0.4 to 7.1]
  Tapis Roulant: number analyzed (Participants) | 2 | 5 | 3
  Tapis Roulant | 0.5 [-5.9 to 6.9] | 1.2 [-1.5 to 3.9] | 5.0 [-7.4 to 17.4]
  Gym Weights: number analyzed (Participants) | 3 | 3 | 5
  Gym Weights | 0.7 [-1.2 to 2.6] | 3.7 [-10.0 to 17.3] | 2.8 [-0.1 to 5.7]
  Exercises at Intervals: number analyzed (Participants) | 4 | 6 | 7
  Exercises at Intervals | 0.8 [-0.8 to 2.3] | 0.0 [0.0 to 0.0] | 2.6 [-0.9 to 6.2]
  General: number analyzed (Participants) | 6 | 22 | 24
  General | 11.2 [3.0 to 19.3] | 5.2 [3.1 to 7.3] | 5.8 [3.4 to 8.2]
  Walk | 3.9 [1.5 to 6.4] | 3.3 [2.2 to 4.4] | 4.7 [2.7 to 6.7]
Statistical Analysis 1: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Running: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.6151, Kruskal-Wallis
Statistical Analysis 2: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Swimming: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.9332, Kruskal-Wallis
Statistical Analysis 3: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Tapis Roulant: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.4726, Kruskal-Wallis
Statistical Analysis 4: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Gym Weights: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.4111, Kruskal-Wallis
Statistical Analysis 5: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Exercises at Intervals: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.0892, Kruskal-Wallis
Statistical Analysis 6: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; General: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.1642, Kruskal-Wallis
Statistical Analysis 7: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Walk: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.7256, Kruskal-Wallis

6. Secondary Outcome: Mean Active Minutes by Intensity (Fairly Active Minutes) for Each Type of Physical Activity Performed by Participants (by Age Categories: 12-17, 18-30, and 31-50 Years) Over the Course of the Study
Description: The number of active minutes by intensity (lightly, fairly, and very active minutes) were obtained at the participant level on a per activity basis as the median of the values collected by the fitness tracker for each activity recorded during the observational period. In this analysis, the means and 95% confidence intervals were calculated using the median fairly active minutes by type of physical activity performed by participants with available data. The physical activities were categorized in the following groups: exercises at intervals, gym weights, running, swimming, tapis roulant, walk, general exercises: other types of physical activity identified by the fitness tracker that are not already included in the above-mentioned categories.
Time Frame: From baseline to study completion (up to 18 months)
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: fairly active minutes per activity
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care:31-50 Years
Number analyzed (Participants) | 6 | 22 | 26
fairly active minutes per activity
  Running: number analyzed (Participants) | 5 | 11 | 8
  Running | 0.0 [0.0 to 0.0] | 1.1 [0.2 to 2.0] | 0.3 [-0.1 to 0.6]
  Swimming: number analyzed (Participants) | 3 | 7 | 8
  Swimming | 1.7 [-5.5 to 8.8] | 6.3 [2.5 to 10.1] | 4.5 [-0.3 to 9.3]
  Tapis Roulant: number analyzed (Participants) | 2 | 5 | 3
  Tapis Roulant | 0.0 [0.0 to 0.0] | 2.3 [0.5 to 4.1] | 1.5 [-2.2 to 5.2]
  Gym Weights: number analyzed (Participants) | 3 | 3 | 5
  Gym Weights | 0.2 [-0.6 to 0.9] | 8.3 [-21.3 to 38.0] | 8.7 [0.1 to 17.3]
  Exercises at Intervals: number analyzed (Participants) | 4 | 6 | 7
  Exercises at Intervals | 1.3 [-2.7 to 5.2] | 0.1 [-0.1 to 0.3] | 0.0 [0.0 to 0.0]
  General: number analyzed (Participants) | 6 | 22 | 24
  General | 13.6 [5.6 to 21.6] | 11.3 [8.4 to 14.2] | 7.9 [3.9 to 11.8]
  Walk | 13.2 [8.0 to 18.3] | 9.8 [7.8 to 11.8] | 9.6 [7.8 to 11.3]
Statistical Analysis 1: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Running: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.0745, Kruskal-Wallis
Statistical Analysis 2: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Swimming: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.2177, Kruskal-Wallis
Statistical Analysis 3: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Tapis Roulant: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.2121, Kruskal-Wallis
Statistical Analysis 4: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Gym weights: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.2336, Kruskal-Wallis
Statistical Analysis 5: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Exercises at intervals: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.4190, Kruskal-Wallis
Statistical Analysis 6: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; General: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.0252, Kruskal-Wallis
Statistical Analysis 7: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care:31-50 Years; Walk: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.2143, Kruskal-Wallis

7. Secondary Outcome: Mean Active Minutes by Intensity (MVPA Minutes) for Each Type of Physical Activity Performed by Participants (by Age Categories: 12-17, 18-30, and 31-50 Years) Over the Course of the Study
Description: The number of active minutes by intensity (lightly, fairly, and very active minutes) were obtained at the participant level on a per activity basis as the median of the values collected by the fitness tracker for each activity recorded during the observational period. The MVPA minutes is the sum of fairly active and very active minutes. In this analysis, the means and 95% confidence intervals were calculated using the median MVPA minutes by type of physical activity performed by participants with available data. The physical activities were categorized in the following groups: exercises at intervals, gym weights, running, swimming, tapis roulant, walk, general exercises: other types of physical activity identified by the fitness tracker that are not already included in the above-mentioned categories.
Time Frame: From baseline to study completion (up to 18 months)
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: MVPA minutes per activity
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care: 31-50 Years
Number analyzed (Participants) | 6 | 22 | 26
MVPA minutes per activity
  Running: number analyzed (Participants) | 5 | 11 | 8
  Running | 4.3 [-4.3 to 12.9] | 36.6 [21.4 to 51.8] | 12.8 [-0.2 to 25.7]
  Swimming: number analyzed (Participants) | 3 | 7 | 8
  Swimming | 2.3 [-7.7 to 12.4] | 14.4 [4.3 to 24.4] | 6.4 [-0.9 to 13.6]
  Tapis Roulant: number analyzed (Participants) | 2 | 5 | 3
  Tapis Roulant | 0 [0 to 0] | 18.8 [0.5 to 37.1] | 17.5 [-34.2 to 69.2]
  Gym weights: number analyzed (Participants) | 3 | 3 | 5
  Gym weights | 5.0 [-16.5 to 26.5] | 49.3 [-56.8 to 155.5] | 29.6 [-9.8 to 69.0]
  Exercise at Intervals: number analyzed (Participants) | 4 | 6 | 7
  Exercise at Intervals | 4.3 [-3.8 to 12.3] | 0.1 [-0.1 to 0.3] | 0 [0 to 0]
  General: number analyzed (Participants) | 6 | 22 | 24
  General | 32.9 [9.5 to 56.3] | 34.3 [23.2 to 45.4] | 26.5 [14.3 to 38.6]
  Walk | 24.2 [15.3 to 33.0] | 33.7 [28.1 to 39.2] | 30.3 [20.7 to 39.8]
Statistical Analysis 1: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Running: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.0085, Kruskal-Wallis
Statistical Analysis 2: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Swimming: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.1098, Kruskal-Wallis
Statistical Analysis 3: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Tapis Roulant: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.2703, Kruskal-Wallis
Statistical Analysis 4: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Gym Weights: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.3366, Kruskal-Wallis
Statistical Analysis 5: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Exercises at Intervals: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.0992, Kruskal-Wallis
Statistical Analysis 6: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; General: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.1194, Kruskal-Wallis
Statistical Analysis 7: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Walk: Comparison among age groups was performed using Kruskal-Wallis test; Test type: Other; p = 0.0549, Kruskal-Wallis

8. Secondary Outcome: Percentage of Participants Who Were Adherent to World Health Organization (WHO) Global Recommendations on Physical Activity for Health Over the Course of the Study
Description: A participant was defined "adherent" to WHO guidelines according to the following algorithm: 12-17 years old: MVPA minutes per day >= 60 minutes. 18-50 years old: Fairly active (moderate) minutes per week >= 150 minutes or very active (vigorous) minutes per week >= 75 minutes or an equivalent combination of fairly and very active minutes (i.e., considering 1 fairly active minute as 0.5 very active minutes). A participant who was adherent to the WHO guidelines according to the above definition was defined as an "active participant", otherwise as a "sedentary participant".
Time Frame: From baseline to study completion (up to 18 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care: 31-50 Years
Number analyzed (Participants) | 6 | 22 | 26
percentage of participants
  Yes (Active Subjects) | 0 | 68.2 | 42.3
  No (Sedentary Subjects) | 100 | 31.8 | 57.7
Statistical Analysis 1: Comparison: Standard of Care: 12-17 Years vs Standard of Care: 18-30 Years vs Standard of Care: 31-50 Years; Comparison among age groups was performed using Chi-squared test; Test type: Other; p = 0.0088, Chi-squared

9. Secondary Outcome: Number of Participants by the Presence of Bleeds (0 vs. ≥1 Bleeds) Over the Course of the Study, Reported Via the ePRO Application
Description: Bleeds that occurred the same day but in different body site were counted separately.
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care:18-30 Years: Participants who were 18-30 years of age with severe or moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
- Standard of Care: 31-50 Years: Participants who were 31- 50 years of age with severe or moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Standard of Care: 12-17 Years | Standard of Care:18-30 Years | Standard of Care: 31-50 Years
Number analyzed (Participants) | 17 | 46 | 40
Participants
  0 Bleeds | 11 | 25 | 22
  1 or More Bleeds | 6 | 21 | 18

10. Secondary Outcome: Number of Participants by the Presence of Bleeds (0 vs. ≥1 Bleeds) Over the Course of the Study According to the Different Types of Bleeds (Spontaneous, Traumatic and Procedure/Surgery Related), Reported Via the ePRO Application
Description: The assessment of bleeds was divided into spontaneous bleeds, traumatic bleeds, and bleeds related to procedure/surgery. Spontaneous bleeds = the occurrence of hemorrhage where neither the participant nor a caregiver could identify a reason. Traumatic bleeds = hemorrhage occurring secondary to an event such as trauma, "strenuous" activity, or "overuse". Bleeds related to procedure/surgery = such as hematomas resulting from any surgeries or invasive procedures.
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months).
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care: 31-50 Years
Number analyzed (Participants) | 17 | 46 | 40
Participants
  Spontaneous Bleed: 0 Bleeds | 15 | 36 | 33
  Spontaneous Bleed: 1 or More Bleeds | 2 | 10 | 7
  Traumatic Bleed: 0 Bleeds | 14 | 28 | 26
  Traumatic Bleed: 1 or More Bleeds | 3 | 18 | 14
  Bleeds Related to Procedures/Surgeries: 0 Bleeds | 17 | 46 | 39
  Bleeds Related to Procedures/Surgeries: 1 or More Bleeds | 0 | 0 | 1

11. Secondary Outcome: Number of Participants by the Presence of Bleeds (0 vs. ≥1 Bleeds) Over the Course of the Study According to the Bleed Sites (Urine, Feces, and Vomit, Joint, Muscle, and Other Bleeds), Reported Via the ePRO Application
Description: Sites of bleeds were defined as urine, faeces, and vomit (three sites grouped together), joint, muscle, and other bleeds.
Time Frame: Baseline and whenever bleeding occured from study initiation to completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care: 12-17 Years | Standard of Care: 18-30 Years | Standard of Care: 31-50 Years
Number analyzed (Participants) | 17 | 46 | 40
Participants
  Urine, Faeces, and Vomit Bleeds: 0 Bleeds | 17 | 45 | 36
  Urine, Faeces, and Vomit Bleeds: 1 or More Bleeds | 0 | 1 | 4
  Joint Bleeds: 0 Bleeds | 13 | 31 | 26
  Joint Bleeds: 1 or More Bleeds | 4 | 15 | 14
  Muscle Bleeds: 0 Bleeds | 15 | 40 | 36
  Muscle Bleeds: 1 or More Bleeds | 2 | 6 | 4
  Other Bleeds: 0 Bleeds | 15 | 40 | 34
  Other Bleeds: 1 or More Bleeds | 2 | 6 | 6

12. Secondary Outcome: Number of Participants by the Type of Regimen Used for Treatment of Haemophilia A Over the Course of the Study
Description: The following types of regimens used to treat haemophilia A are reported here: on-demand (to stop bleeding) and prophylaxis (regular infusions of clotting factor to prevent bleeds). Participants could have received more than one medication.
Time Frame: From baseline to study completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Participants
  Prophylaxis For Haemophilia | 102
  On Demand for Haemophilia | 1

13. Secondary Outcome: Number of Participants by the Product Used for Treatment of Haemophilia A Over the Course of the Study
Description: Participants could have received more than one medication.
Time Frame: From baseline to study completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Participants
  Prophylaxis for Haemophilia: Octocog Alfa | 39
  Prophylaxis for Haemophilia: Efmoroctocog alfa | 25
  Prophylaxis for Haemophilia: Moroctocog Alfa | 8
  Prophylaxis for Haemophilia: Turoctocog Alfa | 8
  Prophylaxis for Haemophilia: Lonoctocog Alfa | 6
  Prophylaxis for Haemophilia: Rurioctocog Alfa Pegol | 6
  Prophylaxis for Haemophilia: Damoctocog Alfa Pegol | 3
  Prophylaxis for Haemophilia: Simoctocog Alfa | 3
  Prophylaxis for Haemophilia: Turoctocog Alfa Pegol | 3
  Prophylaxis for Haemophilia: Factor VIII (Antihaemophilic Factor) | 2
  Prophylaxis for Haemophilia: Factor VIII, Recombinant | 1
  Prophylaxis for Haemophilia: Emicizumab | 17
  Prophylaxis for Haemophilia: Desmopressin | 1
  Prophylaxis for Haemophilia: Tranexamic Acid | 2
  On Demand for Haemophilia: Octocog Alfa | 1

14. Secondary Outcome: Number of Participants Who Switched to a New Approved Drug for Treatment of Haemophilia A by the Product Used
Description: Participants could have received more than one medication.
Time Frame: From baseline to the time of switch to a new therapy (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Participants
  Turoctocog Alfa Pegol | 7
  Damoctocog Alfa Pegol | 3
  Rurioctocog Alfa Pegol | 3
  Emicizumab | 8

15. Secondary Outcome: Number of Treated Bleeds Over the Course of the Study
Description: An event was considered a treated bleed if coagulation factors were administered to treat signs or symptoms of bleeding (e.g., pain, swelling, etc.).
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker. Overall number of bleeds analyzed=number of bleeds during analysis at given timepoint.
Measure: Number; unit: number of treated bleeds
Units Other Than Participants: Bleeds
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Number analyzed (Bleeds) | 129
number of treated bleeds | 94

16. Secondary Outcome: Number of Bleeds Treated With Each Type of Treatment for Bleeding (Haemostatic Treatment, Treatment for Pain)
Description: as for outcome 15
Time Frame: From baseline to whenever bleeding occurred (up to 18 months)
Population: as for outcome 15
Measure: Number; unit: number of treated bleeds
Units Other Than Participants: Treated bleeds
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Number analyzed (Treated bleeds) | 94
number of treated bleeds
  Haemostatic Treatment | 93
  Treatment for Pain | 1

17. Secondary Outcome: Duration of Treatment for Bleeding Over the Course of the Study
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Median (Full Range); unit: days
Units Other Than Participants: Treated bleeds
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Number analyzed (Treated bleeds) | 94
days | 2.0 [1 to 18]

18. Secondary Outcome: Number of Bleeds Treated With Each Route of Administration Over the Course of the Study
Description: Number of bleeds treated by intravenous, subcutaneous, intramuscular, nasal, ophthalmic, oral, rectal, and other routes of administration are reported here.
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months)
Population: as for outcome 15
Measure: Number; unit: number of treated bleeds
Units Other Than Participants: Treated bleeds
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Number analyzed (Treated bleeds) | 94
number of treated bleeds
  Intravenous | 90
  Subcutaneous | 0
  Intramuscular | 0
  Nasal | 0
  Ophthalmic | 0
  Oral | 4
  Rectal | 0
  Others | 0

19. Secondary Outcome: Number of Bleeds Which Needed to Receive a Transfusion
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months)
Population: as for outcome 15
Measure: Number; unit: number of bleeds
Units Other Than Participants: Bleeds
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Number analyzed (Bleeds) | 129
number of bleeds | 0

20. Secondary Outcome: Number of Bleeds Which Needed to Administer an Additional Hemostatic Therapy
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months)
Population: as for outcome 15
Measure: Number; unit: number of bleeds
Units Other Than Participants: Bleeds
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Number analyzed (Bleeds) | 129
number of bleeds | 4

21. Secondary Outcome: Number of Bleeds With Adherence to Treatment Regimen for Haemophilia A in the Week Preceding the Bleeding
Description: The adherence to the treatment regimen for haemophilia A was analyzed as the number of bleeds with an answer equal to "Yes" and "My therapeutic plan does not include any treatment in the last week" in the week preceding the bleeding.
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months)
Population: as for outcome 15
Measure: Number; unit: Number of bleeds
Units Other Than Participants: Bleeds
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Number analyzed (Bleeds) | 129
Number of bleeds | 77

22. Secondary Outcome: Number of Participants Who Were Adherent to the Treatment Regimen for Haemophilia A Over the Course of the Study by Adherence Category (<80% vs. ≥80% of Study Weeks)
Description: The adherence to the treatment regimen for haemophilia A was analyzed as the number of participants with <80% or ≥80% of weeks on study with "Yes" and "My therapeutic plan does not include any treatment in the last week" over the total number of weeks reported via the ePRO. Missing data from some weeks was treated as "No". The total number of weeks on study for each participant was derived as (End of study date - Baseline date + 1) / 7.
Time Frame: From baseline to study completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker. A total of 4 participants had missing data and were excluded from this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 99
Participants
  Adherence <80% of Weeks | 72
  Adherence ≥80% of Weeks | 27

23. Secondary Outcome: Number of Participants by the Product of Concomitant Medications Taken to Control Pain Over the Course of the Study
Description: Participants could have received more than one medication.
Time Frame: Baseline and every 3 months until study completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 103
Participants
  Etoricoxib | 5
  Paracetamol | 4

24. Secondary Outcome: Pain Intensity, as Reported by Participants Using a Visual Analogue Scale
Description: Participants reported the intensity of pain in their main joints (elbow, knee, ankle) by marking on a visual analogue scale (VAS), a horizontal line 100 millimeters (mm) in length, anchored by word descriptors at each end, where the left extreme means "No pain = 0" while the right extreme means "Worst Pain Imaginable = 100". The VAS score is the distance (in mm) from the left end of the line to the point where the participant marks crossed the line. VAS scale was submitted to the participants every month during the study.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at given timepoints.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 100
scores on a scale
  Baseline | 14.24 [10.09 to 18.39]
  Month 1: number analyzed (Participants) | 82
  Month 1 | 18.38 [13.5 to 23.26]
  Month 2: number analyzed (Participants) | 78
  Month 2 | 16.91 [11.97 to 21.85]
  Month 3: number analyzed (Participants) | 79
  Month 3 | 17.53 [12.77 to 22.28]
  Month 4: number analyzed (Participants) | 79
  Month 4 | 21.77 [16.10 to 27.44]
  Month 5: number analyzed (Participants) | 71
  Month 5 | 18.76 [13.37 to 24.15]
  Month 6: number analyzed (Participants) | 75
  Month 6 | 18.98 [13.99 to 23.97]
  Month 7: number analyzed (Participants) | 63
  Month 7 | 19.89 [14.19 to 25.59]
  Month 8: number analyzed (Participants) | 65
  Month 8 | 17.85 [12.17 to 23.54]
  Month 9: number analyzed (Participants) | 55
  Month 9 | 17.58 [11.8 to 23.36]
  Month 10: number analyzed (Participants) | 66
  Month 10 | 18.20 [12.75 to 23.65]
  Month 11: number analyzed (Participants) | 55
  Month 11 | 20.26 [14.31 to 26.22]
  Month 12: number analyzed (Participants) | 60
  Month 12 | 19.85 [13.88 to 25.82]
  Month 13: number analyzed (Participants) | 4
  Month 13 | 29.50 [-18.53 to 77.53]
  Month 14: number analyzed (Participants) | 5
  Month 14 | 21.40 [-2.85 to 45.65]
  Month 15: number analyzed (Participants) | 4
  Month 15 | 20.75 [-2.97 to 44.47]
  Month 16: number analyzed (Participants) | 2
  Month 16 | 12.50 [-146.33 to 171.33]
  Month 17: number analyzed (Participants) | 2
  Month 17 | 15 [-175.59 to 205.59]
  Month 18: number analyzed (Participants) | 2
  Month 18 | 1.00 [-11.71 to 13.71]

25. Secondary Outcome: Health-Related Quality of Life (HRQoL): European Quality of Life-5 Dimensions (EQ-5D-5L) Health State Utility Index Score Over Time
Description: The EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L includes five levels of severity in each of the five EuroQol-5D dimensions and the EQ VAS. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each dimension having 5 levels (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems). Response options are measured with a 5-point Likert scale. The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state and lower score indicate worse health state. EQ-5D-5L questionnaire was submitted to the participants every 3 month from baseline during the study.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 100
scores on a scale
  Baseline | 0.93 [0.91 to 0.94]
  Month 1: number analyzed (Participants) | 1
  Month 1 | 0.89 [NA to NA] — Due to low number of participants, upper and lower limits of 95% CI could not be calculated.
  Month 2: number analyzed (Participants) | 0
  Month 3: number analyzed (Participants) | 78
  Month 3 | 0.90 [0.88 to 0.93]
  Month 4: number analyzed (Participants) | 8
  Month 4 | 0.94 [0.90 to 0.98]
  Month 5: number analyzed (Participants) | 2
  Month 5 | 0.94 [0.11 to 1.76]
  Month 6: number analyzed (Participants) | 76
  Month 6 | 0.90 [0.88 to 0.92]
  Month 7: number analyzed (Participants) | 5
  Month 7 | 0.92 [0.83 to 1.01]
  Month 8: number analyzed (Participants) | 49
  Month 8 | 0.93 [0.90 to 0.95]
  Month 9: number analyzed (Participants) | 25
  Month 9 | 0.88 [0.85 to 0.91]
  Month 10: number analyzed (Participants) | 4
  Month 10 | 0.80 [0.62 to 0.97]
  Month 11: number analyzed (Participants) | 52
  Month 11 | 0.90 [0.87 to 0.92]
  Month 12: number analyzed (Participants) | 25
  Month 12 | 0.92 [0.89 to 0.96]
  Month 13: number analyzed (Participants) | 1
  Month 13 | 0.62 [NA to NA] — Due to low number of participants, upper and lower limits of 95% CI could not be calculated.
  Month 14: number analyzed (Participants) | 4
  Month 14 | 0.86 [0.79 to 0.93]
  Month 15: number analyzed (Participants) | 1
  Month 15 | 0.85 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 16: number analyzed (Participants) | 0
  Month 17: number analyzed (Participants) | 2
  Month 17 | 0.90 [-0.33 to 2.14]
  Month 18: number analyzed (Participants) | 1
  Month 18 | 0.92 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.

26. Secondary Outcome: Health Status Measured Over Time, as Reported by Participants Using EQ-5D VAS Score
Description: The EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and the other section is an evaluation of the overall health status using VAS. The VAS records the respondent's self-rated health on a 20 centimeter (cm) vertical VAS from 0 to 100 on how good or bad their health is at assessment; 0 means the worst health imaginable, and 100 means the best health imaginable.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 100
scores on a scale
  Baseline | 81.9 [77.8 to 86]
  Month 1: number analyzed (Participants) | 1
  Month 1 | 81.0 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.
  Month 2: number analyzed (Participants) | 0
  Month 3: number analyzed (Participants) | 78
  Month 3 | 80.6 [76.2 to 85.0]
  Month 4: number analyzed (Participants) | 8
  Month 4 | 86.0 [74.4 to 97.6]
  Month 5: number analyzed (Participants) | 2
  Month 5 | 83.5 [-75.3 to 242.3]
  Month 6: number analyzed (Participants) | 76
  Month 6 | 75.8 [70.1 to 81.4]
  Month 7: number analyzed (Participants) | 5
  Month 7 | 64 [29.6 to 98.4]
  Month 8: number analyzed (Participants) | 49
  Month 8 | 78.4 [71.3 to 85.6]
  Month 9: number analyzed (Participants) | 25
  Month 9 | 73.3 [63.1 to 83.5]
  Month 10: number analyzed (Participants) | 4
  Month 10 | 72.5 [40 to 105]
  Month 11: number analyzed (Participants) | 52
  Month 11 | 75.3 [68.6 to 82.1]
  Month 12: number analyzed (Participants) | 25
  Month 12 | 69.6 [55.5 to 83.7]
  Month 13: number analyzed (Participants) | 1
  Month 13 | 65 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.
  Month 14: number analyzed (Participants) | 4
  Month 14 | 83.3 [56.7 to 109.8]
  Month 15: number analyzed (Participants) | 1
  Month 15 | 75 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.
  Month 16: number analyzed (Participants) | 0
  Month 17: number analyzed (Participants) | 2
  Month 17 | 85 [-105.6 to 275.6]
  Month 18: number analyzed (Participants) | 1
  Month 18 | 97 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.

27. Secondary Outcome: Haemophilia Joint Health Score (HJHS) Total Score Over Time
Description: The HJHS is an instrument developed to measure joint health status and to identify early signs of joint disease in children. This tool assesses joints most commonly affected by bleeding (knees, ankles, and elbows). Each of the 6 joints is assessed across 8 domains (Swelling, Duration of Swelling, Atrophy, Crepitus, Flexion Loss, Extension Loss, Pain, and Strength), and a Total Score is calculated as the sum of all joint domain scores. The score range is from 0 to 124 points (a score of 0 indicates no joint damage). A higher score indicates higher joint damage.
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Standard of Care for Haemophilia: Participants with severe or moderate Haemophilia A without inhibitors against Factor VIII, receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Standard of Care for Haemophilia
Number analyzed (Participants) | 102
scores on a scale
  Baseline | 10 [7.2 to 12.7]
  Month 6: number analyzed (Participants) | 20
  Month 6 | 13.7 [3.5 to 23.8]
  Month 12: number analyzed (Participants) | 52
  Month 12 | 12.5 [7.4 to 17.6]

28. Secondary Outcome: Mean Body Mass Index (BMI) Over Time
Time Frame: Baseline, Months 3, 6, 9, 12, 15 and 18
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: kilogram per square meter (kg/m2)
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 101
kilogram per square meter (kg/m2)
  Baseline | 23.34 [22.64 to 24.05]
  Month 3: number analyzed (Participants) | 12
  Month 3 | 23.56 [22.26 to 24.86]
  Month 6: number analyzed (Participants) | 30
  Month 6 | 23.42 [22.02 to 24.82]
  Month 9: number analyzed (Participants) | 11
  Month 9 | 23.76 [21.31 to 26.21]
  Month 12: number analyzed (Participants) | 39
  Month 12 | 22.98 [21.88 to 24.07]
  Month 15: number analyzed (Participants) | 0
  Month 18: number analyzed (Participants) | 0

29. Secondary Outcome: Yearly Rate of Days Away From School or Work for Participants
Description: The number of days away from school or work (participant) was analyzed every month as a continuous variable. The yearly rate was derived on a per participant basis as the proportion between the total number of days away from school and/or work and the duration of the study (derived as end of study date - baseline date + 1) multiplied by 365.25.
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: days/year
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 96
days/year | 0 [0 to 57]

30. Secondary Outcome: Yearly Rate of Days Away From Work for Parent/Caregiver
Description: The number of days away from work was analyzed every month as a continuous variable. The yearly rate was derived on a per participant (for parents and caregivers) basis as the proportion between the total number of days away from work and duration of the study (derived as end of study date - baseline date + 1) multiplied by 365.25.
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: as for outcome 29
Measure: Median (Full Range); unit: days/year
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 96
days/year | 0 [0 to 57]

31. Secondary Outcome: Yearly Rate of Hospitalization Days
Description: The yearly rate was derived on a per participant basis as the proportion between the total number of hospitalization days and the duration of the study (derived as end of study date - baseline date + 1) multiplied by 365.25.
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: as for outcome 29
Measure: Median (Full Range); unit: days/year
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 96
days/year | 0.0 [0 to 15.6]

32. Secondary Outcome: Age of Possible Early Retirement of Caregiver, as Reported by Caregivers in a Questionnaire
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: as for outcome 29
Measure: Mean (95% Confidence Interval); unit: years
Arm/Group | Standard of Care for Haemophilia A
Number analyzed (Participants) | 8
years | 57.8 [38.1 to 77.4]

33. Secondary Outcome: Number of Active Versus Sedentary Participants by the Severity (Moderate or Severe) of Haemophilia A
Description: Participants who were adherent to the WHO guidelines for physical activity according to the below definition were defined as an "active participant", otherwise as a "sedentary participant". A participant was defined "adherent" to WHO guidelines according to the following algorithm: 12-17 years old: MVPA minutes per day >= 60 minutes. 18-50 years old: Fairly active (moderate) minutes per week >= 150 minutes or Very active (vigorous) minutes per week >= 75 minutes or an equivalent combination of fairly and very active minutes (i.e., considering 1 fairly active minute as 0.5 very active minutes). The participants were classified as 'Active' or 'Sedentary' based on data collected from baseline till the end of the study.
Time Frame: From baseline up to study completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Groups:
- Moderate Haemophilia A: Participants with moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
- Severe Haemophilia A: Participants with severe Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 97
Participants
  Sedentary Participants | 3 | 54
  Active Participants | 3 | 34
  Unknown | 0 | 9

34. Secondary Outcome: Annualized Bleeding Rates (ABR) in Active Versus Sedentary Participants
Description: The annualized bleeding rate was derived as follows: total number of bleeds/total follow-up (person-year), where the individual's study duration was given by ([end of study date-baseline date +1] divided by 365.25). ABR was reported in active and sedentary participants. A participant who was adherent to the WHO guidelines for physical activity according to the below definition was defined as an "active participant", otherwise as a "sedentary participant". WHO guidelines for adherence: 12-17 years old: MVPA minutes per day >= 60 minutes. 18-50 years old: Fairly active (moderate) minutes per week >= 150 minutes or Very active (vigorous) minutes per week >= 75 minutes or an equivalent combination of fairly and very active minutes (i.e., considering 1 fairly active minute as 0.5 very active minutes).
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: rate of bleeds per person-year
Groups:
- Sedentary Participants: Participants with severe or moderate Haemophilia A without inhibitors against Factor VIII, who classified as 'Sedentary' per WHO physical activity guideline, receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
- Active Participants: Participants with severe or moderate Haemophilia A without inhibitors against Factor VIII, who classified as 'Active' per WHO physical activity guideline, receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
rate of bleeds per person-year | 1.945 [1.481 to 2.509] | 1.384 [0.974 to 1.907]

35. Secondary Outcome: Pain Intensity in Active Versus Sedentary Participants, as Reported by Participants Using a Visual Analogue Scale
Description: Participants reported intensity of pain in their main joints (elbow, knee, ankle) by marking on a VAS, a horizontal line 100 mm in length, anchored by word descriptors at each end, where the left extreme means "No pain = 0" while right extreme means "Worst Pain Imaginable = 100". VAS score is the distance (in mm) from left end of the line to the point where participant marks crossed the line. A participant who was adherent to WHO guidelines for physical activity according to the below definition was defined as an "active participant", otherwise as a "sedentary participant". WHO guidelines for adherence: 12-17 years old: MVPA minutes per day ≥60 minutes. 18-50 years old: Fairly active (moderate) minutes per week ≥150 minutes or Very active (vigorous) minutes per week ≥75 minutes or an equivalent combination of fairly and very active minutes (i.e., considering 1 fairly active minute as 0.5 very active minutes). VAS scale was submitted to the participants every month during the study.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: Evaluable population included all enrolled participants with at least 6 valid months of physical activity evaluations during the study. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
scores on a scale
  Baseline: number analyzed (Participants) | 28 | 25
  Baseline | 17.86 [8.84 to 26.87] | 14.12 [4.80 to 23.44]
  Month 1: number analyzed (Participants) | 24 | 26
  Month 1 | 21.29 [11.95 to 30.63] | 15.73 [7.03 to 24.43]
  Month 2: number analyzed (Participants) | 25 | 24
  Month 2 | 18.32 [10.83 to 25.81] | 16.75 [6.89 to 26.61]
  Month 3: number analyzed (Participants) | 25 | 23
  Month 3 | 22.80 [14.38 to 31.22] | 17.17 [7.82 to 26.53]
  Month 4: number analyzed (Participants) | 25 | 23
  Month 4 | 27.56 [17.11 to 38.01] | 24.22 [11.83 to 36.61]
  Month 5: number analyzed (Participants) | 25 | 23
  Month 5 | 23.28 [13.28 to 33.28] | 20 [8.69 to 31.31]
  Month 6: number analyzed (Participants) | 23 | 24
  Month 6 | 24.09 [13.13 to 35.04] | 20.67 [10.73 to 30.61]
  Month 7: number analyzed (Participants) | 21 | 23
  Month 7 | 22.52 [12.16 to 32.89] | 20.78 [10.90 to 30.67]
  Month 8: number analyzed (Participants) | 22 | 20
  Month 8 | 22.02 [10.81 to 33.23] | 19.98 [8.34 to 31.61]
  Month 9: number analyzed (Participants) | 23 | 18
  Month 9 | 17.80 [7.43 to 28.18] | 24.81 [13.64 to 35.97]
  Month 10: number analyzed (Participants) | 22 | 22
  Month 10 | 20.16 [8.92 to 31.40] | 20.98 [11.65 to 30.30]
  Month 11: number analyzed (Participants) | 23 | 22
  Month 11 | 20.72 [10.23 to 31.21] | 21.09 [11.97 to 30.21]
  Month 12: number analyzed (Participants) | 19 | 17
  Month 12 | 22.68 [10.94 to 34.43] | 25 [12.11 to 37.89]
  Month 13: number analyzed (Participants) | 2 | 2
  Month 13 | 7.50 [-87.80 to 102.80] | 51.50 [-183.56 to 286.56]
  Month 14: number analyzed (Participants) | 3 | 1
  Month 14 | 8.33 [-10.64 to 27.31] | 33 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 15: number analyzed (Participants) | 3 | 1
  Month 15 | 16.67 [-21.28 to 54.61] | 33 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 16: number analyzed (Participants) | 2 | 0
  Month 16 | 12.50 [-146.33 to 171.33] |
  Month 17: number analyzed (Participants) | 2 | 0
  Month 17 | 15 [-175.59 to 205.59] |
  Month 18: number analyzed (Participants) | 2 | 0
  Month 18 | 1 [-11.71 to 13.71] |

36. Secondary Outcome: Number of Active Versus Sedentary Participants by the Product of Concomitant Medications Taken to Control Pain Over the Course of the Study
Description: A participant who was adherent to the WHO guidelines for physical activity according to the below definition was defined as an "active participant", otherwise as a "sedentary participant". WHO guidelines for adherence: 12-17 years old: MVPA minutes per day >= 60 minutes. 18-50 years old: Fairly active (moderate) minutes per week >= 150 minutes or Very active (vigorous) minutes per week >= 75 minutes or an equivalent combination of fairly and very active minutes (i.e., considering 1 fairly active minute as 0.5 very active minutes). Participants can have received more than one medication.
Time Frame: Baseline and every 3 months until study completion (up to 18 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Sedentary Participants: Participants with severe or moderate Haemophilia A without inhibitors against Factor VIII, who classified as 'Sedentary' per WHO physical activities guideline, receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
- Active Participants: Participants with severe or moderate Haemophilia A without inhibitors against Factor VIII, who classified as 'Active' per WHO physical activities guideline, receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
Participants
  Etoricoxib | 2 | 2
  Paracetamol | 1 | 2

37. Secondary Outcome: Number of Active Versus Sedentary Participants by the Type of Regimen Used for Treatment of Haemophilia A Over the Course of the Study
Description: The following types of regimens used to treat haemophilia A are reported here: on-demand (to stop bleeding) and prophylaxis (regular infusions of clotting factor to prevent bleeds). A participant who was adherent to the WHO guidelines for physical activity according to the below definition was defined as an "active participant", otherwise as a "sedentary participant". WHO guidelines for adherence: 12-17 years old: MVPA minutes per day >= 60 minutes. 18-50 years old: Fairly active (moderate) minutes per week >= 150 minutes or Very active (vigorous) minutes per week >= 75 minutes or an equivalent combination of fairly and very active minutes (i.e., considering 1 fairly active minute as 0.5 very active minutes). Participants can have received more than one medication.
Time Frame: From baseline to study completion (up to 18 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
Participants
  Prophylaxis for Haemophilia | 28 | 25
  On Demand for Haemophilia | 0 | 1

38. Secondary Outcome: Number of Active Versus Sedentary Participants by the Product Used for Treatment of Haemophilia A Over the Course of the Study
Description: A participant who was adherent to the WHO guidelines for physical activity according to the below definition was defined as an "active participant", otherwise as a "sedentary participant". WHO guidelines for adherence: 12-17 years old: MVPA minutes per day >= 60 minutes. 18-50 years old: Fairly active (moderate) minutes per week >= 150 minutes or Very active (vigorous) minutes per week >= 75 minutes or an equivalent combination of fairly and very active minutes (i.e., considering 1 fairly active minute as 0.5 very active minutes).
Time Frame: From baseline to study completion (up to 18 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
Participants
  Prophylaxis for Haemophilia: Octocog Alfa | 8 | 10
  Prophylaxis for Haemophilia: Efmoroctocog Alfa | 8 | 7
  Prophylaxis for Haemophilia: Moroctocog Alfa | 3 | 2
  Prophylaxis for Haemophilia: Turoctocog Alfa | 1 | 3
  Prophylaxis for Haemophilia: Lonoctocog Alfa | 3 | 0
  Prophylaxis for Haemophilia: Rurioctocog Alfa Pegol | 2 | 1
  Prophylaxis for Haemophilia: Simoctocog Alfa | 3 | 0
  Prophylaxis for Haemophilia: Turoctocog Alfa Pegol | 1 | 2
  Prophylaxis for Haemophilia: Damoctocog Alfa Pegol | 0 | 1
  Prophylaxis for Haemophilia: Factor VIII (Antihemophilic Factor) | 0 | 1
  Prophylaxis for Haemophilia: Emicizumab | 6 | 3
  Prophylaxis for Haemophilia: Tranexamic Acid | 1 | 1
  On Demand for Haemophilia: Octocog Alfa | 0 | 1

39. Secondary Outcome: Number of Active Versus Sedentary Participants Who Switched to a New Approved Drug for Treatment of Haemophilia A by the Product Used
Description: as for outcome 38
Time Frame: From baseline to the time of switch to a new therapy (up to 18 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
Participants
  Turoctocog Alfa Pegol | 1 | 4
  Damoctocog Alfa Pegol | 1 | 1
  Rurioctocog Alfa Pegol | 1 | 0
  Emicizumab | 5 | 0

40. Secondary Outcome: HRQoL: EQ-5D-5L Health State Utility Index Score Over Time for Active Versus Sedentary Participants
Description: EQ-5D-5L is a standardized measure of health status developed by EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L includes five levels of severity in each of five EuroQol-5D dimensions and EQ VAS. Descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each dimension having 5 levels (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems). Response options are measured with a 5-point Likert scale. 5D-5L systems are converted into a single index utility score between 0-1, where higher score indicates a better health state and lower score indicate worse health state. A participant who was adherent to WHO guidelines for physical activity was defined as an "active participant", otherwise as a "sedentary participant". EQ-5D-5L questionnaire was submitted to participants every 3 month from baseline during the study.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: Evaluable population included all enrolled participants with at least 6 valid months of physical activity evaluations during the study. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at given timepoints.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 25
scores on a scale
  Baseline | 0.90 [0.86 to 0.94] | 0.93 [0.90 to 0.95]
  Month 1: number analyzed (Participants) | 0 | 1
  Month 1 |  | 0.89 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 2: number analyzed (Participants) | 0 | 0
  Month 3: number analyzed (Participants) | 25 | 23
  Month 3 | 0.89 [0.84 to 0.93] | 0.90 [0.86 to 0.94]
  Month 4: number analyzed (Participants) | 2 | 1
  Month 4 | 0.95 [0.33 to 1.57] | 1 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 5: number analyzed (Participants) | 0 | 0
  Month 6: number analyzed (Participants) | 24 | 24
  Month 6 | 0.87 [0.81 to 0.92] | 0.90 [0.87 to 0.93]
  Month 7: number analyzed (Participants) | 2 | 2
  Month 7 | 0.87 [0.74 to 0.99] | 0.94 [0.11 to 1.76]
  Month 8: number analyzed (Participants) | 17 | 16
  Month 8 | 0.9 [0.86 to 0.94] | 0.91 [0.87 to 0.95]
  Month 9: number analyzed (Participants) | 10 | 9
  Month 9 | 0.85 [0.80 to 0.91] | 0.88 [0.81 to 0.94]
  Month 10: number analyzed (Participants) | 0 | 0
  Month 11: number analyzed (Participants) | 22 | 22
  Month 11 | 0.89 [0.85 to 0.94] | 0.89 [0.85 to 0.93]
  Month 12: number analyzed (Participants) | 5 | 4
  Month 12 | 0.86 [0.74 to 0.98] | 0.97 [0.88 to 1.06]
  Month 13: number analyzed (Participants) | 0 | 1
  Month 13 |  | 0.62 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 14: number analyzed (Participants) | 2 | 1
  Month 14 | 0.89 [0.38 to 1.39] | 0.86 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated..
  Month 15: number analyzed (Participants) | 1 | 0
  Month 15 | 0.85 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated. |
  Month 16: number analyzed (Participants) | 0 | 0
  Month 17: number analyzed (Participants) | 2 | 0
  Month 17 | 0.90 [-0.33 to 2.14] |
  Month 18: number analyzed (Participants) | 1 | 0
  Month 18 | 0.92 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated. |

41. Secondary Outcome: Health Status Measured Over Time, as Reported by Participants Using EQ-5D VAS Score in Active Versus Sedentary Participants
Description: The EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities pain/discomfort, anxiety/depression) and the other section is an evaluation of the overall health status using VAS. The VAS records the respondent's self-rated health on a 20 centimeter (cm) vertical VAS from 0 to 100 on how good or bad their health is at assessment; 0 means the worst health imaginable, and 100 means the best health imaginable. A participant who was adherent to the WHO guidelines for physical activity was defined as an "active participant", otherwise as a "sedentary participant".
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: as for outcome 40
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 25
scores on a scale
  Baseline | 79.9 [72.9 to 86.8] | 78.1 [66.7 to 89.5]
  Month 1: number analyzed (Participants) | 0 | 1
  Month 1 |  | 81.0 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 2: number analyzed (Participants) | 0 | 0
  Month 3: number analyzed (Participants) | 25 | 23
  Month 3 | 76.9 [68.7 to 85.1] | 81.8 [74.3 to 89.3]
  Month 4: number analyzed (Participants) | 2 | 1
  Month 4 | 80.0 [-174.1 to 334.1] | 97.0 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 5: number analyzed (Participants) | 0 | 0
  Month 6: number analyzed (Participants) | 24 | 24
  Month 6 | 73.1 [62.8 to 83.4] | 76.1 [67.3 to 84.9]
  Month 7: number analyzed (Participants) | 2 | 2
  Month 7 | 62.5 [30.7 to 94.3] | 55.0 [-389.7 to 499.7]
  Month 8: number analyzed (Participants) | 17 | 16
  Month 8 | 80.2 [70.2 to 90.2] | 79.1 [66.8 to 91.5]
  Month 9: number analyzed (Participants) | 10 | 9
  Month 9 | 70.7 [53 to 88.4] | 67.0 [44.1 to 89.9]
  Month 10: number analyzed (Participants) | 0 | 0
  Month 11: number analyzed (Participants) | 22 | 22
  Month 11 | 81.7 [74.5 to 88.9] | 66.7 [53.7 to 79.7]
  Month 12: number analyzed (Participants) | 5 | 4
  Month 12 | 47.8 [7.2 to 88.4] | 89.3 [79.5 to 99.0]
  Month 13: number analyzed (Participants) | 0 | 1
  Month 13 |  | 65.0 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 14: number analyzed (Participants) | 2 | 1
  Month 14 | 97.5 [65.7 to 129.3] | 67.0 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated.
  Month 15: number analyzed (Participants) | 1 | 0
  Month 15 | 75 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated. |
  Month 16: number analyzed (Participants) | 0 | 0
  Month 17: number analyzed (Participants) | 2 | 0
  Month 17 | 85.0 [-105.6 to 275.6] |
  Month 18: number analyzed (Participants) | 1 | 0
  Month 18 | 97 [NA to NA] — Since only one participants was evaluated upper and lower limit of 95% CI could not be calculated. |

42. Secondary Outcome: HJHS Total Score for Active Versus Sedentary Participants Over Time
Description: as for outcome 27
Time Frame: Baseline, Months 6 and 12
Population: Evaluable population included all enrolled participants with at least 6 valid months of physical activity evaluations during the study. Number analyzed is the number of participants with data available for analysis at given timepoint.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
scores on a scale
  Baseline | 11.8 [5.1 to 18.4] | 12.1 [6.2 to 18.0]
  Month 6: number analyzed (Participants) | 6 | 6
  Month 6 | 29.3 [-7.3 to 66.0] | 8.7 [3.0 to 14.4]
  Month 12: number analyzed (Participants) | 18 | 14
  Month 12 | 17.3 [4.8 to 29.9] | 15.0 [5.4 to 24.6]

43. Secondary Outcome: Yearly Rate of Number of Days Away From School/Work for Active Versus Sedentary Participants
Description: as for outcome 29
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: days/year
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
days/year | 0.0 [0 to 57] | 0.0 [0 to 12]

44. Secondary Outcome: Yearly Rate of Number of Days Away From Work for Active Versus Sedentary Participant's Parents or Caregivers
Description: The number of days away from work was analyzed every month as a continuous variable. The yearly rate was derived on a per participant (for parents/caregivers) basis as the proportion between the total number of days away from work and the duration of the study (derived as end of study date - baseline date + 1) multiplied by 365.25.
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: days/year
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
days/year | 0.0 [0 to 57] | 0.0 [0 to 4]

45. Secondary Outcome: Yearly Rate of Number of Hospitalization Days for Active Versus Sedentary Participants
Description: as for outcome 31
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 28 | 26
days | 0 [0.0 to 5.0] | 0 [0.0 to 0.9]

46. Secondary Outcome: Annualized Bleeding Rates in Active Versus Sedentary Participants by the Severity (Moderate Versus Severe) of Haemophilia A
Description: The annualized bleeding rate was derived as follows: total number of bleeds/total follow-up (person-year), where the individual's study duration was given by ([end of study date-baseline date +1] divided by 365.25). A participant who was adherent to the WHO guidelines for physical activity was defined as an "active participant", otherwise as a "sedentary participant". Participants were classified for disease severity at baseline: severe (Factor VIII activity <1%) or moderate (Factor VIII activity between ≥1% and ≤2%) haemophilia A.
Time Frame: Baseline and whenever bleeding occurred from study initiation to completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker. Overall number of participants analyzed is the number of participants with available physical activities data in ITT population for sedentary and active participants.
Measure: Mean (95% Confidence Interval); unit: rate of bleeds per person-year
Groups:
- Active Participants: Participants severe or moderate Haemophilia A without inhibitors against Factor VIII, who classified as 'Active' per WHO physical activity guideline, receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Sedentary Participants | Active Participants
Number analyzed (Participants) | 57 | 37
rate of bleeds per person-year
  Moderate Haemophilia: number analyzed (Participants) | 3 | 3
  Moderate Haemophilia | 0.368 [0.009 to 2.049] | 2.536 [1.095 to 4.998]
  Severe Haemophilia: number analyzed (Participants) | 54 | 34
  Severe Haemophilia | 1.517 [1.212 to 1.876] | 1.035 [0.717 to 1.446]

47. Secondary Outcome: Pain Intensity in Participants With Moderate Versus Severe Haemophilia A, as Reported by Participants Using a Visual Analogue Scale
Description: Participants reported the intensity of pain in their main joints (elbow, knee, ankle) by marking on a VAS, a horizontal line 100 mm in length, anchored by word descriptors at each end, where the left extreme means "No pain = 0" while the right extreme means "Worst Pain Imaginable = 100". The VAS score is the distance (in mm) from the left end of the line to the point where the participant marks crossed the line. VAS scale was submitted to the participants every month during the study.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17 and 18
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at given timepoint.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 94
scores on a scale
  Baseline | 23.33 [-5.34 to 52.01] | 13.66 [9.46 to 17.86]
  Month 1: number analyzed (Participants) | 6 | 76
  Month 1 | 23.67 [-8.87 to 56.20] | 17.96 [13.03 to 22.90]
  Month 2: number analyzed (Participants) | 5 | 73
  Month 2 | 19.20 [-19.80 to 58.20] | 16.75 [11.76 to 21.75]
  Month 3: number analyzed (Participants) | 5 | 74
  Month 3 | 21.00 [-14.78 to 56.78] | 17.29 [12.46 to 22.12]
  Month 4: number analyzed (Participants) | 5 | 74
  Month 4 | 29.00 [-9.87 to 67.87] | 21.28 [15.48 to 27.09]
  Month 5: number analyzed (Participants) | 5 | 66
  Month 5 | 26.20 [-10.17 to 62.57] | 18.20 [12.69 to 23.70]
  Month 6: number analyzed (Participants) | 5 | 70
  Month 6 | 26.40 [-1.01 to 53.81] | 18.45 [13.27 to 23.63]
  Month 7: number analyzed (Participants) | 4 | 59
  Month 7 | 28.75 [-15.94 to 73.44] | 19.29 [13.46 to 25.12]
  Month 8: number analyzed (Participants) | 4 | 61
  Month 8 | 27.63 [-17.84 to 73.09] | 17.21 [11.41 to 23.02]
  Month 9: number analyzed (Participants) | 5 | 50
  Month 9 | 17.00 [-13.29 to 47.29] | 17.64 [11.58 to 23.70]
  Month 10: number analyzed (Participants) | 4 | 62
  Month 10 | 19.38 [7.30 to 31.45] | 18.12 [12.33 to 23.91]
  Month 11: number analyzed (Participants) | 4 | 51
  Month 11 | 11.50 [0.75 to 22.25] | 20.95 [14.57 to 27.33]
  Month 12: number analyzed (Participants) | 3 | 57
  Month 12 | 19.33 [-3.75 to 42.41] | 19.88 [13.60 to 26.16]
  Month 13: number analyzed (Participants) | 1 | 3
  Month 13 | 70.00 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated. | 16.00 [-25.04 to 57.04]
  Month 14: number analyzed (Participants) | 0 | 5
  Month 14 |  | 21.40 [-2.85 to 45.65]
  Month 15: number analyzed (Participants) | 0 | 4
  Month 15 |  | 20.75 [-2.97 to 44.47]
  Month 16: number analyzed (Participants) | 0 | 2
  Month 16 |  | 12.50 [-146.33 to 171.33]
  Month 17: number analyzed (Participants) | 0 | 2
  Month 17 |  | 15.00 [-175.59 to 205.59]
  Month 18: number analyzed (Participants) | 0 | 2
  Month 18 |  | 1.00 [-11.71 to 13.71]

48. Secondary Outcome: Number of Participants With Moderate Versus Severe Haemophilia A by the Product of Concomitant Medications Taken to Control Pain Over the Course of the Study
Description: Participants could have received more than one medication.
Time Frame: Baseline and every 3 months until study completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 97
Participants
  Etoricoxib | 0 | 5
  Paracetamol | 0 | 4

49. Secondary Outcome: Number of Participants With Moderate Versus Severe Haemophilia A by the Type of Regimen Used for Treatment of Haemophilia A Over the Course of the Study
Description: as for outcome 12
Time Frame: From baseline to study completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Groups:
- Moderate Haemophilia: Participants with moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Moderate Haemophilia | Severe Haemophilia A
Number analyzed (Participants) | 6 | 97
Participants
  Prophylaxis for Haemophilia | 5 | 97
  On Demand for Haemophilia | 1 | 0

50. Secondary Outcome: Number of Participants With Moderate Versus Severe Haemophilia A by the Product Used for Treatment of Haemophilia A
Description: Participants could have received more than one medication.
Time Frame: From baseline to study completion (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 97
Participants
  Prophylaxis; Octocog Alfa | 1 | 38
  Prophylaxis; Efmoroctocog Alfa | 2 | 23
  Prophylaxis; Moroctocog Alfa | 1 | 7
  Prophylaxis; Turoctocog Alfa | 0 | 8
  Prophylaxis; Lonoctocog Alfa | 0 | 6
  Prophylaxis; Rurioctocog Alfa Pegol | 0 | 6
  Prophylaxis; Damoctocog Alfa Pegol | 0 | 3
  Prophylaxis; Simoctocog Alfa | 1 | 2
  Prophylaxis; Turoctocog Alfa Pegol | 0 | 3
  Prophylaxis; Factor VIII (Antihaemophilic Factor) | 0 | 2
  Prophylaxis; Factor VIII, Recombinant | 0 | 1
  Prophylaxis; Emicizumab | 0 | 17
  Prophylaxis; Desmopressin | 0 | 1
  Prophylaxis; Tranexamic Acid | 1 | 1
  On Demand; Octocog Alfa | 1 | 0

51. Secondary Outcome: Number of Participants With Moderate Versus Severe Haemophilia A Who Switched to a New Approved Drug for Treatment of Haemophilia A by the Product Used
Description: Participants could have received more than one medication.
Time Frame: From baseline to the time of switch to a new therapy (up to 18 months)
Population: ITT population included all enrolled participants who received the ePRO application and the fitness tracker.
Measure: Count of Participants; unit: Participants
Groups:
- Moderate Haemophilia A: Participants who were 12-17 years of Participants with moderate Haemophilia A without inhibitors against Factor VIII receiving standard of care treatment, independently of participation in the current study, according to clinician's independent therapeutic decision were enrolled for a maximum observation period of 18 months.
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 97
Participants
  Turoctocog Alfa Pegol | 2 | 5
  Damoctocog Alfa Pegol | 0 | 3
  Rurioctocog Alfa Pegol | 0 | 3
  Emicizumab | 0 | 8

52. Secondary Outcome: HRQoL: EQ-5D-5L Health State Utility Index Score Over Time Moderate Versus Severe Haemophilia A
Description: as for outcome 25
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: as for outcome 47
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Moderate Haemophilia | Severe Haemophilia A
Number analyzed (Participants) | 6 | 94
scores on a scale
  Baseline | 0.92 [0.84 to 1.0] | 0.93 [0.91 to 0.94]
  Month 1: number analyzed (Participants) | 0 | 1
  Month 1 |  | 0.89 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.
  Month 2: number analyzed (Participants) | 0 | 0
  Month 3: number analyzed (Participants) | 5 | 73
  Month 3 | 0.88 [0.67 to 1.09] | 0.90 [0.88 to 0.93]
  Month 4: number analyzed (Participants) | 1 | 7
  Month 4 | 0.90 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated. | 0.95 [0.90 to 0.99]
  Month 5: number analyzed (Participants) | 0 | 2
  Month 5 |  | 0.94 [0.11 to 1.76]
  Month 6: number analyzed (Participants) | 5 | 71
  Month 6 | 0.92 [0.79 to 1.05] | 0.90 [0.87 to 0.92]
  Month 7: number analyzed (Participants) | 0 | 5
  Month 7 |  | 0.92 [0.83 to 1.01]
  Month 8: number analyzed (Participants) | 2 | 47
  Month 8 | 0.91 [0.79 to 1.03] | 0.93 [0.90 to 0.95]
  Month 9: number analyzed (Participants) | 3 | 22
  Month 9 | 0.83 [0.49 to 1.18] | 0.88 [0.85 to 0.91]
  Month 10: number analyzed (Participants) | 0 | 4
  Month 10 |  | 0.80 [0.62 to 0.97]
  Month 11: number analyzed (Participants) | 4 | 48
  Month 11 | 0.93 [0.85 to 1.01] | 0.90 [0.87 to 0.92]
  Month 12: number analyzed (Participants) | 0 | 25
  Month 12 |  | 0.92 [0.89 to 0.96]
  Month 13: number analyzed (Participants) | 1 | 0
  Month 13 | 0.62 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated. |
  Month 14: number analyzed (Participants) | 0 | 4
  Month 14 |  | 0.86 [0.79 to 0.93]
  Month 15: number analyzed (Participants) | 0 | 1
  Month 15 |  | 0.85 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.
  Month 16: number analyzed (Participants) | 0 | 0
  Month 17: number analyzed (Participants) | 0 | 2
  Month 17 |  | 0.90 [-0.33 to 2.14]
  Month 18: number analyzed (Participants) | 0 | 1
  Month 18 |  | 0.92 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.

53. Secondary Outcome: Health Status Measured Over Time, as Reported by Participants Using EQ-5D VAS Score in Participants With Moderate Versus Severe Haemophilia A
Description: The EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and the other section is an evaluation of the overall health status using VAS. The VAS records the respondent's self-rated health on a 20 cm vertical VAS from 0 to 100 on how good or bad their health is at assessment; 0 means the worst health imaginable, and 100 means the best health imaginable.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: as for outcome 47
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 94
scores on a scale
  Baseline | 88.3 [72.9 to 103.8] | 81.5 [77.2 to 85.8]
  Month 1: number analyzed (Participants) | 0 | 1
  Month 1 |  | 81.0 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.
  Month 2: number analyzed (Participants) | 0 | 0
  Month 3: number analyzed (Participants) | 5 | 73
  Month 3 | 81.2 [54.6 to 107.8] | 80.5 [76.0 to 85.1]
  Month 4: number analyzed (Participants) | 1 | 7
  Month 4 | 75.0 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated. | 87.6 [74.4 to 100.7]
  Month 5: number analyzed (Participants) | 0 | 2
  Month 5 |  | 83.5 [-75.3 to 242.3]
  Month 6: number analyzed (Participants) | 5 | 71
  Month 6 | 84.4 [71.8 to 97.0] | 75.1 [69.2 to 81.1]
  Month 7: number analyzed (Participants) | 0 | 5
  Month 7 |  | 64.0 [29.6 to 98.4]
  Month 8: number analyzed (Participants) | 2 | 47
  Month 8 | 48 [-358.6 to 454.6] | 79.7 [72.8 to 86.7]
  Month 9: number analyzed (Participants) | 3 | 22
  Month 9 | 82.3 [45.0 to 119.7] | 72.0 [60.6 to 83.5]
  Month 10: number analyzed (Participants) | 0 | 4
  Month 10 |  | 72.5 [40.0 to 105.0]
  Month 11: number analyzed (Participants) | 4 | 48
  Month 11 | 73.5 [21.0 to 126.0] | 75.5 [68.5 to 82.4]
  Month 12: number analyzed (Participants) | 0 | 25
  Month 12 |  | 69.6 [55.5 to 83.7]
  Month 13: number analyzed (Participants) | 1 | 0
  Month 13 | 65.0 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated. |
  Month 14: number analyzed (Participants) | 0 | 4
  Month 14 |  | 83.3 [56.7 to 109.8]
  Month 15: number analyzed (Participants) | 0 | 1
  Month 15 |  | 75.0 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.
  Month 16: number analyzed (Participants) | 0 | 0
  Month 17: number analyzed (Participants) | 0 | 2
  Month 17 |  | 85.0 [-105.6 to 275.6]
  Month 18: number analyzed (Participants) | 0 | 1
  Month 18 |  | 97.0 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated.

54. Secondary Outcome: HJHS Total Score for Participants With Moderate Versus Severe Haemophilia A
Description: The HJHS is an instrument developed to measure joint health status and to identify early signs of joint disease in children. This tool assesses joints most commonly affected by bleeding (knees, ankles, and elbows). Each of the 6 joints is assessed across 8 domains (Swelling, Duration of Swelling, Atrophy, Crepitus, Flexion Loss, Extension Loss, Pain, and Strength), and a Total Score is calculated as the sum of all joint domain scores. The total score range is from 0 to 124 points (a score of 0 indicates no joint damage). A higher score indicates higher joint damage.
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 96
scores on a scale
  Baseline | 8.3 [-1.1 to 17.8] | 10.1 [7.2 to 12.9]
  Month 6: number analyzed (Participants) | 1 | 19
  Month 6 | 20.0 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated. | 13.3 [2.6 to 24]
  Month 12: number analyzed (Participants) | 1 | 51
  Month 12 | 0.0 [NA to NA] — Since only one participant was evaluated, upper and lower limit of 95% CI could not be calculated. | 12.8 [7.6 to 17.9]

55. Secondary Outcome: Yearly Rate of Days Away From School for Participants With Moderate Versus Severe Haemophilia A
Description: as for outcome 29
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: as for outcome 29
Measure: Median (Full Range); unit: days/year
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 90
days/year | 0.0 [0 to 5] | 0.0 [0 to 57]

56. Secondary Outcome: Yearly Rate of Days Away From Work for Parents/Caregivers of Participants With Moderate Versus Severe Haemophilia A
Description: as for outcome 44
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: as for outcome 29
Measure: Median (Full Range); unit: days/year
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 90
days/year | 0.0 [0 to 0] | 0 [0 to 57]

57. Secondary Outcome: Yearly Rate of Hospitalization Days for Participants With Moderate Versus Severe Haemophilia A
Description: as for outcome 31
Time Frame: Baseline and every month until study completion (up to 18 months)
Population: as for outcome 29
Measure: Median (Full Range); unit: days/year
Arm/Group | Moderate Haemophilia A | Severe Haemophilia A
Number analyzed (Participants) | 6 | 90
days/year | 0 [0.0 to 0.0] | 0 [0.0 to 15.6]

ADVERSE EVENTS:
Time Frame: No adverse event data were collected during this study.
Description: As pre-specified in the protocol for this non-interventional study, no adverse event data were actively collected during the study.
Arm/Group | Standard of Care for Haemophilia A
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT04165135/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04165135/SAP_001.pdf